CLINICAL TRIAL: NCT02915198
Title: CSP #2002 - Investigation of Metformin in Pre-Diabetes on Atherosclerotic Cardiovascular OuTcomes (VA-IMPACT)
Brief Title: Investigation of Metformin in Pre-Diabetes on Atherosclerotic Cardiovascular OuTcomes
Acronym: VA-IMPACT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2002
Record Dates: First submitted 2016-09-13; First posted 2016-09-26 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prediabetic State; Atherosclerosis; Metformin
Keywords: Metformin; Atherosclerosis; Prediabetic State; Hemoglobin A, Glycosylated; Coronary Artery Disease; Peripheral Arterial Disease; Cerebrovascular Disorders
MeSH Terms: conditions — Prediabetic State; Atherosclerosis; Coronary Artery Disease; Peripheral Arterial Disease; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Participants receive initial treatment with metformin XR 500 mg 1 tablet daily, with stepwise titration to a maximum dose of 2000 mg (4 tablets) daily.
  Interventions: Drug: Metformin XR
- Placebo (Placebo Comparator): Participants receive initial treatment with 1 tablet daily of placebo (for metformin XR), with stepwise titration to a maximum of 4 tablets daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin XR — The study medication dose may be increased by a step-wise fashion up to a maximum of 4 tablets per day.
  Arms: Metformin
Drug: Placebo — For patients < 80 years of age at the time of a study visit, and with most recent eGFR 45 mL/min/1.73 m2, study medication dose may be increased in a stepwise fashion to a maximum of 4 tablets daily, corresponding to metformin XR 2000 mg or matching placebo.
  For patients 80 years of age or with most recent 30 eGFR < 45 mL/min/1.73 m2, the maximum dose of study medication is 2 tablets daily, corresponding to metformin XR 1000 mg or matching placebo
  Arms: Placebo

SUMMARY:
This research will help us to learn if the medicine called metformin reduces the risk of death, heart attacks, and/or strokes in Veterans who have pre-diabetes and heart or blood vessel problems.

DETAILED DESCRIPTION:
CSP #2002 is a multicenter, prospective, randomized, double blind, secondary prevention trial to test the hypothesis that treatment with metformin, compared with placebo, reduces mortality and cardiovascular morbidity in Veterans with pre-diabetes and established atherosclerotic cardiovascular disease. Qualifying patients have pre-diabetes defined by HbA1c, fasting blood glucose, or oral glucose tolerance test criteria; clinically evident coronary, cerebrovascular, or peripheral arterial atherosclerotic cardiovascular disease; and estimated glomerular filtration rate of at least 45 mL/min/1.73 m2; and do not fulfill any exclusion criteria. Patients who are eligible and agree to participate are randomly assigned to treatment with metformin XR (titrated to a maximum dose of 2000 mg daily based on safety and tolerability) or matching placebo. All patients receive counseling on therapeutic lifestyle recommendations.

CSP #2002 had a Pilot Phase trial from 2/2019 to 1/2021 and was approved for the full-scale trial, with Full-scale study launch in 04/2023.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-diabetes: This condition is fulfilled by HbA1c of at least 5.7%, but less than 6.5%; or two measurements of fasting plasma glucose (on separate days) of 100-125 mg/dL; or a 2-hour plasma glucose level of 140-199 mg/dL following a 75 g glucose load oral glucose tolerance test.
2. Established atherosclerotic cardiovascular disease: Qualifying participants must have evidence of atherosclerotic disease in at least one of the following vascular beds: coronary, cerebrovascular, or peripheral arterial circulation.

Coronary artery disease is fulfilled by at least one of (1), (2), or (3):

1. History of myocardial infarction at least one month prior to randomization.
2. History of percutaneous coronary intervention or coronary artery bypass surgery at least one month prior to randomization.
3. Angiographic evidence of coronary stenosis of at least 50% in at least two major epicardial coronary arteries.

Cerebrovascular disease is fulfilled by at least one of criteria (1) through (4):

1. Documented prior ischemic stroke (at least one month prior to randomization),
2. Carotid artery stenosis 50% and history of transient ischemic attack or transient ischemic visual symptoms attributable to the identified lesion(s),
3. Asymptomatic carotid stenosis of at least 70% luminal diameter,
4. History of carotid revascularization (surgical or catheter-based).

Peripheral arterial disease: Fulfilled by at least one of the following:

1. History of aorto-iliac or peripheral artery intervention (surgical or catheter based) for limb ischemia, or amputation for limb ischemia,
2. Symptoms of intermittent claudication with ankle:brachial index less than or equal to 0.85.

3. Renal function: Estimated glomerular filtration rate at least 45 mL/min/1.73 m2.

4. Informed consent has been fully executed, and participant agrees to study procedures.

Exclusion Criteria:

1. Treatment with metformin or other anti-diabetic medication within 12 months of randomization. Note: In the absence of a diagnosis of diabetes, inpatient treatment with insulin or treatment with an SGLT2 inhibitor (e.g., for heart failure) or a GLP-1 receptor agonist (e.g., for obesity) is not exclusionary.
2. Treatment with systemic glucocorticoids within 3 months of randomization
3. Fasting plasma glucose greater than 130 mg/dL measured between screening and randomization visits, or any plasma glucose 180 mg/dL or HbA1c 7.0% measured within 12 months of randomization.
4. Total CO2 below the local laboratory lower limit of normal on most recent blood chemistry panel
5. Current treatment with cimetidine, vandetanib, or a systemic treatment with a carbonic anhydrase inhibitor.
6. Cirrhosis, active hepatitis, or jaundice at time of randomization, or total bilirubin > 2 times upper limit of normal
7. Binge or heavy alcohol consumption within 6 months of randomization
8. Severe anemia (hemoglobin < 10 g/dL)
9. Prior history of intolerance to metformin
10. Myocardial infarction, coronary revascularization procedure, or stroke within 1 month of randomization
11. Uncontrolled hypertension at screening assessment (systolic blood pressure 180 mm Hg or diastolic blood pressure 110 mm Hg
12. Acute or decompensated congestive heart failure
13. Expected survival less than study duration
14. Participants considered to be unable, unwilling, or unreliable to meet protocol requirements
15. Impaired decision-making capacity, defined by any history of dementia or cognitive impairment
16. Concurrent participation in another research study involving a randomized comparison of drug or device treatments, unless specifically excepted.
17. Pregnant, intent to become pregnant during the trial, or lactating
18. Women of childbearing potential who are not using a highly effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7410 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2029-09-28 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Time in days to death, non-fatal myocardial infarction, stroke, hospitalization for unstable angina, or symptom-driven coronary revascularization | through study completion, an average of 4.5 years
  The primary outcome measure is the time to first occurrence of death, non-fatal myocardial infarction or stroke, hospitalization for unstable angina with objective evidence of acute myocardial ischemia, or coronary revascularization driven by acute or progressive symptoms.

SECONDARY OUTCOMES:
Time in days to Cardiovascular Outcomes | through study completion, an average of 4.5 years
  * Time to first occurrence of death, myocardial infarction, or stroke
  * Time to first occurrence of a primary endpoint event, peripheral arterial disease event, or hospitalization for congestive heart failure
  * Cumulative incidence of all components of the primary endpoint, including recurrent or multiple events in the same participant
  * Cumulative incidence and time to first occurrence of each component of the primary outcome measure, peripheral arterial disease events, and hospitalization for congestive heart failure
Time in days to Oncologic Outcome | through study completion, an average of 4.5 years
  Time to new or recurrent diagnosis of a malignancy or death from a malignancy
Time in days to Diabetes Outcome | through study completion, an average of 4.5 years
  Time to new diagnosis of type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Gregory G. Schwartz, PhD MD, Study Chair — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (40):
- United States (40):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Pacific Islands Health Care System, Honolulu, HI, Honolulu, Hawaii
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Lexington VA Medical Center, Lexington, KY, Lexington, Kentucky
  - Rehabilitation R&D Service, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - Huntington VA Medical Center, Huntington, WV, Huntington, West Virginia
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No